CLINICAL TRIAL: NCT04681261
Title: Evaluation of Occupational Balance, Fear and Agoraphobia in Adults
Brief Title: Occupational Balance, Fear and Agoraphobia
Acronym: OB
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İnal, principal investigator, Hacettepe University
Other Study IDs: 2020/185
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: this study is not an intervention study — this study is not an intervention study

SUMMARY:
This study was planned to investigate occupational balance, fear of Covid-19 and agoraphobia in adults during the Covid-19 pandemic.

DETAILED DESCRIPTION:
During the Covid-19 pandemic, the occupational balance of individuals change and the sedentary activities preferences, that pose a risk for health, increase.The outbreak also produced effects such as fear of sickness and death in addition to changing daily life and work routines, occupational balance and social participation. This study was planned to investigate occupational balance, fear of Covid-19 and agoraphobia in adults during the Covid-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

between 19-65 years of age

Exclusion Criteria:

<19 years and >65 years old

Ages: 19 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult individuals
Sampling Method: Probability Sample
Enrollment: 699 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Occupational Balance Questionnaire | 3 months
  The Occupational Balance Questionnaire (OBQ) is a scale that measures self-rated OB in different dimensions. 11 item in the scale is scored on a 4-point scale from 'strongly disagree' to 'strongly agree'. The total score is obtained by summing the individual items and ranges from 0 to 33, with higher scores indicating higher OB.

CONTACTS AND LOCATIONS:
Overall Officials: Özgü İnal, Principal Investigator — Trakya University
Locations (1):
- Özgü İnal, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No